CLINICAL TRIAL: NCT00628069
Title: The Effect of Bench-model Training in Cognitive Learning in the Operating Room
Status: Completed | Type: Observational
Sponsor: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Khalid Syed, Orthopedic Surgeon, The Physicians' Services Incorporated Foundation
Other Study IDs: 07-43
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Sensitivity Training Groups
Keywords: Orthopedics; bone fixation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1: performers who will participate in the training sessions.
- Assistants: Assisants-paired with the performers and will be allowed to assists only, without the opportunity to practice the technical skills related to the task.

SUMMARY:
Based on the motor learning theories, it is hypothesized that bench-model training will allow junior residents to be more interactive than trainees lacking similar active hands-on training.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in first or second year of their residency from a variety of division

Exclusion Criteria:

* Residents from higher year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents enrolled in first or second year from a variety of divisions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to show that bench model testing not only improves the technical skill of the student but that it also influences the student's ability to learn the didactic information and decision-making. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Syed, MD, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada